CLINICAL TRIAL: NCT03698409
Title: Onabotulinumtoxin Type A Reconstitution With Preserved Versus Preservative-free Saline in Chronic Migraine. A Randomized, Double-blind Trial.
Brief Title: Onabotulinumtoxin Type A Reconstitution With Preserved Versus Preservative-free Saline in Chronic Migraine.
Acronym: B-RECON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Awss Zidan, MD, Clinical Instructor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1318956
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Chronic Migraine, Headache
Keywords: Migraine; Onabotulinumtoxin A; Botox; Reconstitution; Saline
MeSH Terms: conditions — Headache; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox in preservative-free saline (No Intervention): OnabotulinumtoxinA (Botox) 200u will be reconstituted using 4 ml of preservative-free saline, as recommended by the manufacturer. 155-195 u of Onabotulinumtoxin A (Botox) will be injected in subjects with chronic migraine, consistent with FDA-approval indications, following the standard injection protocol (31 sites)
- Botox in preserved saline (Active Comparator): OnabotulinumtoxinA (Botox) 200u will be reconstituted using 4 ml of preservative saline (i.e. bacteriostatic saline). 155-195 u of Onabotulinumtoxin A (Botox) will be injected in subjects with chronic migraine, consistent with FDA-approval indications, following the standard injection protocol (31 sites).
  Interventions: Drug: Preserved saline in reconstitution of Botox

INTERVENTIONS:
Drug: Preserved saline in reconstitution of Botox — The intervention consists of using 4 ml of preserved saline for the reconstitution of OnabotuliniumtoxinA prior to its use in subjects with chronic migraine.
  Other Names: Bacteriostatic saline
  Arms: Botox in preserved saline

SUMMARY:
A growing body of literature on the cosmetic use of OnabotulinumtoxinA has suggested that the use of preserved saline exerts a local anesthetic effect, and reduces the procedure discomfort when used in reconstitution in lieu of preservative-free saline. However, this has never been studied in chronic migraine.

While reducing discomfort is a desirable target in all procedures, it has a special importance in the use of OnabotulinumtoxinA for chronic migraine due to the numerous injection locations each session (31 sites) and the ubiquity of scalp tenderness in this population. In addition, the pain during procedure is a known migraine trigger for many of these patients.

We hypothesize that preserved saline (known as bacteriostatic saline) produces lower procedure-related discomfort when used as a dissolving solution for OnabotulinumtoxinA in individuals with chronic migraine as opposed to using preservative-free saline.

In addition, we hypothesize that reduction of procedure-relate pain during the injections will also result in reduced migraine/headache attacks in the week immediately following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of chronic migraine receiving FDA-approved treatment with OnabotulinumtoxinA injection as per standard protocol. Standard protocol consists of 31 injection sites, with total dose ranging from 155 u to 195u.

Exclusion Criteria:

* Subjects whom OnabotulinumtoxinA injections deviate from standard protocol for any reason, such as head/neck infection, head deformity, recent surgery…etc.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the headache clinic of SUNY Upstate Medical University which is a tertiary care center in central New York. Two of the authors performed the randomization through a simulated "coin flipper" website (www.random.org). Following the randomization, same authors prepared the syringes. Two different authors performed the injections.
Period: Overall Study
Arm/Group | Botox in Preservative-free Saline | Botox in Preserved Saline
Started | 39 | 29
Completed | 39 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox in Preservative-free Saline | Botox in Preserved Saline | Total
Number analyzed (Participants) | 39 | 29 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.5) | 43 (14.3) | 43 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 9 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 39 | 29 | 68

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Scale
Description: Difference in verbal pain scale (0 to 10, 0 indicates no pain, and 10 indicates most severe pain)
Time Frame: Immediately after intervention, an average of 2 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Botox in Preservative-free Saline | Botox in Preserved Saline
Number analyzed (Participants) | 39 | 29
score on a scale | 5.3 [4.8 to 6.1] | 3.3 [2.5 to 4.1]

2. Secondary Outcome: Headache-day Frequency
Description: Difference in headache-days in the first week following the procedure
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Botox in Preservative-free Saline | Botox in Preserved Saline
Number analyzed (Participants) | 39 | 29
days | 4.6 (2.3) | 4.1 (1.7)

ADVERSE EVENTS:
Time Frame: up to 7 days
Arm/Group | Botox in Preservative-free Saline | Botox in Preserved Saline
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/29
Other Adverse Events (participants affected / at risk) | 0/39 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT03698409/Prot_SAP_001.pdf